CLINICAL TRIAL: NCT00677885
Title: Measurement of P-Glycoprotein Function in Alzheimer Disease, Parkinson Disease, and Frontotemporal Dementia Using Positron Emission Tomography
Brief Title: P-glycoprotein Function in Brain Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080124; 08-M-0124
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2014-08-25

CONDITIONS: Alzheimer Disease; Parkinson Disease; Frontotemporal Lobar Degeneration
Keywords: Alzheimer Disease; Parkinson's Disease; Frontotemporal Dementia; PET Imaging; AD; Parkinson Disease; PD
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Frontotemporal Lobar Degeneration; Frontotemporal Dementia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will measure the function of a protein called P-glycoprotein (P-gp), which is found at the blood-brain barrier, a membrane that normally prevents toxic material from entering the brain. Impaired P-gp function may allow toxins to enter the brain and cause some people to develop certain brain diseases.

Healthy subjects and people with Alzheimer s disease, Parkinson s disease or frontotemporal dementia who are 35 years of age or older and in overall good health may be eligible for this study.

Participants undergo the following procedures during three outpatient visits to the NIH Clinical Center:

* Medical history, psychological evaluation, physical examination and blood and urine tests, including tests for illegal and addictive drugs.
* PET scan: This test uses small amounts of a radioactive chemical called a tracer that labels active areas of the brain so the activity can be seen with a special camera. Before starting the scan, a catheter (plastic tube) is placed in a vein in the arm to inject the tracer. The subject lies on the scanner bed, with a special mask fitted to the head and attached to the bed to help keep the head still during the scan so the images obtained are clear. A brief initial scan is done to calibrate the scanner. Then, a radioactive tracer called [(15)O]H(2)O is injected into the catheter and the PET camera takes pictures of blood flow to the brain for about 60 seconds. Next, another tracer, [(11)C]dLop, is injected into the catheter and pictures are taken for about 2 hours to determine how much of this tracer is allowed to enter the brain.
* Magnetic resonance imaging (MRI): This procedure is done within 1 year (before or after) the PET scan. MRI uses a magnetic field and radio waves to produce images of the brain. For this procedure, the patient lies on a table that can slide in and out of the scanner (a tube-like device), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scan.

DETAILED DESCRIPTION:
Objective

Alzheimer disease (AD), Parkinson disease (PD), and frontotemporal dementia (FTD) are associated with the accumulation of neurotoxic material in the brain. Potentially toxic material is normally restricted from the brain by P-glycoprotein, a transporter protein expressed by endothelial cells at the blood-brain barrier. Disruption of the blood-brain barrier has been reported in animal models of AD, PD, and FTD, and specific dysfunction of P-gp has been linked to AD and PD pathology. Therefore, P-gp may be protective against certain neurodegenerative diseases, and P-gp dysfunction may be a risk factor for developing AD, PD, or FTD.

Positron emission tomography (PET) imaging can measure P-gp function. If P-gp function is abnormal, a radiolabeled P-gp substrate will cross the blood-brain barrier and enter the brain. Intact P-gp function, on the other hand, will prevent the substrate from entering the brain. If P-gp dysfunction is a risk factor for developing AD, PD, or FTD, then patients with these diseases should have more radiolabeled substrate in the brain than healthy controls.

We have developed a novel radioligand, [(11)C]N-desmethyl-loperamide [(11)C]dLop), which is a P-gp substrate. Our goal is to use PET imaging with [(11)C]dLop to see if P-gp function is reduced in AD, PD, and FTD.

Study population

In this protocol, we wish to evaluate 15 patients with AD, 15 patients with PD, 15 patients with FTD, and 15 healthy volunteers.

Design

Subjects will undergo screening with a history, physical exam, ECG, and blood and urine laboratory testing. Subjects will receive a dedicated brain PET with [(11)C]dLop and a brain MRI. Since [11C]dLop uptake is influenced by blood flow, a [(15)O]H2O PET scan will be performed to determine flow to the brain.

Outcome measures

Our outcome measure will be the amount of [(11)C]dLop uptake in the brain in AD, PD, and FTD patients and in healthy controls. Brain uptake will be measured as the percent standardized uptake value (%SUV). Percent SUV reflects the measured brain radioactivity after [(11)C]dLop injection, corrected for patient weight and the injected dose of [(11)C]dLop. As an exploratory outcome measure, we also will correct brain uptake for cerebral blood flow. Blood flow will be determined using [(15)O]H2O PET.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with the diagnosis of probable Alzheimer disease, Parkinson disease, or frontotemporal dementia. All patients must either meet capacity criteria to consent to research, or be able to assign a surrogate decision-maker who is able to consent to research on the subject s behalf.
* Healthy volunteers.

EXCLUSION CRITERIA:

* Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam.
* Laboratory tests with clinically significant abnormalities.
* Subjects on blood-thinning medications, having coagulation disorders, or clinically significant abnormal blood clotting test (PT/PTT).
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure, including that from this protocol, would exceed the guidelines set by the Radiation Safety Committee (RSC).
* Pregnancy or breast feeding.
* Positive result on urine screen for illicit drugs.
* Subjects who cannot lie on their back for extended periods of time.
* History of neurological disease other than Alzheimer disease, Parkinson disease, or frontotemporal dementia.
* Subjects who have a cardiac pacemaker or metal in their body.
* Subjects taking cyclosporine A.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05-09; Study Completion 2014-08-25

PRIMARY OUTCOMES:
P-gp function in AD, PD, and FTD patients and in healthy volunteers. P-gp function will be determined by calculating the brain uptake of [11C]dLop

SECONDARY OUTCOMES:
Comparing P-gp function with the severity of disease

CONTACTS AND LOCATIONS:
Overall Officials: William C Kreisl, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hochman JH, Pudvah N, Qiu J, Yamazaki M, Tang C, Lin JH, Prueksaritanont T. Interactions of human P-glycoprotein with simvastatin, simvastatin acid, and atorvastatin. Pharm Res. 2004 Sep;21(9):1686-91. doi: 10.1023/b:pham.0000041466.84653.8c. PMID 15497697
- [Background] Mahar Doan KM, Humphreys JE, Webster LO, Wring SA, Shampine LJ, Serabjit-Singh CJ, Adkison KK, Polli JW. Passive permeability and P-glycoprotein-mediated efflux differentiate central nervous system (CNS) and non-CNS marketed drugs. J Pharmacol Exp Ther. 2002 Dec;303(3):1029-37. doi: 10.1124/jpet.102.039255. PMID 12438524
- [Background] Schwab D, Fischer H, Tabatabaei A, Poli S, Huwyler J. Comparison of in vitro P-glycoprotein screening assays: recommendations for their use in drug discovery. J Med Chem. 2003 Apr 24;46(9):1716-25. doi: 10.1021/jm021012t. PMID 12699389